CLINICAL TRIAL: NCT03289858
Title: Does the Use of Liposomal Bupivacaine Decrease Narcotic Requirements in Geriatric Hip Fractures? A Randomized, Double Blinded Control Trial
Brief Title: Randomized Controlled Trial for Exparel Hip Fracture
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Orthopaedic Trauma Association (Other); University of Kentucky (Other)
Responsible Party: Principal Investigator, Eric Swart, Eric F. Swart, MD, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H00013594
Record Dates: First submitted 2017-09-08; First posted 2017-09-21 (Actual); Results first posted 2020-02-25 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Exparel (Liposomal Bupivacaine) (Experimental): Exparel (liposomal bupivacaine) is FDA approved, with a labeled indication of "single-dose infiltration into the surgical site to produce postsurgical analgesia."
  Interventions: Drug: Exparel
- Saline Control (Placebo Comparator): Saline Solution (Sodium Chloride)
  Interventions: Drug: Sodium Chloride

INTERVENTIONS:
Drug: Exparel — Subcutaneous injection at conclusion of surgical fixation of hip fracture
  Other Names: Liposomal Bupivacaine
  Arms: Exparel (Liposomal Bupivacaine)
Drug: Sodium Chloride — Saline Injection
  Other Names: Saline
  Arms: Saline Control

SUMMARY:
This is a prospective, randomized study looking at the effect that a long-acting local anesthetic has on pain control in patients having surgery for hip fractures. The investigators are conducting the study to see if that reduces the amount of pain medicine needed after surgery, and if it reduces other medical complications after surgery.

DETAILED DESCRIPTION:
Osteoporotic fragility fractures of the hip are common in the geriatric population, are increasing in frequency, and represent a growing social and economic burden. Pain control after surgical treatment is an area of growing interest, as improvement in post-injury pain is often an important indication for surgical treatment of hip fractures.

Typically a mainstay of post-operative pain control, the use of opiates has come under increasing scrutiny, as it has been shown to be associated with delirium, respiratory depression, and even may even lead to addiction or abuse in the medically frail geriatric population. These concerns have led to efforts to minimize the use of post-operative opiates in hip fracture patients. In that context, a treatment that could reduce the necessity of post-op narcotics while still improving pain control would be potentially valuable.

There has been growing interest in the use of long-acting local anesthetics for improving pain control in orthopaedics, particularly in the elective total joint arthroplasty population. Studies have shown that arthroplasty patients receiving long-acting local anesthetics have decreased opiate requirements, reduced length of stay, and lower costs. Although well-demonstrated in the elective arthroplasty population, the effects of long-acting local anesthetics have yet to be demonstrated in the hip fracture population. Given that these fractures frequently occur in medically frail patients with multiple comorbidities, in whom post-operative confusion and delirium are relatively common, there is the potential for treatments that decrease opiate requirements to demonstrate substantial medical and economic benefits.

Exparel (liposomal bupivacaine) and long-acting local anesthetics have been used extensively in hip replacement surgery and have not been shown to be associated with any increased risks. In the case of patients with displaced femoral neck fractures treated with arthroplasty, the surgical techniques are identical to those being used in this study. Exparel has also been used in trauma surgery as well as foot and ankle surgery without any increased described risks, although its use explicitly in hip fractures has not been published. However, the PI has trained in other medical centers where Exparel is routinely used in hip fracture patients without any identified increased risks or complications, but there is a paucity of data on this subject, which is the rationale for this study.

The investigators hypothesize that in patients with osteoporotic fragility fractures of the hip, patients receiving intraoperative long-acting local anesthetics will have decreased pain and decreased post-operative opiate requirements, leading to less delirium and decreased hospital resource utilization during their index hospitalization.

The goal is to conduct a multi-center prospective randomized control trial to determine if liposomal bupivacaine is superior to standard of care by addressing the below separate but related aims:

1. Determine the effectiveness of Exparel to reduce narcotic requirements and pain post operatively after hip fracture treatment. Excess narcotic use in the elderly population is associated with a host of complications often magnified by polypharmacy, including in hospital delirium, increased length of stay, nausea, constipation, urinary retention, respiratory depression and others. Decreasing narcotic usage in this group of patients following hip fracture can possibly reduce such complications. Patients will receive standard of care medical treatment and be randomized to intra-operative Exparel vs. placebo injections. Opioid requirements, complications, pain score, and length of stay will be assessed in the post-operative period. Hypothesis: The investigators hypothesize that total morphine requirements and pain scores will be decreased in this group following the administration of exparel in the geriatric hip fracture fracture population.
2. Determine the effectiveness of Exparel to reduce delirium in post-operative hip fracture patients. In hospital delirium in elderly patients is associated with poor outcomes, including prolonged length of stay, poor participation in rehabilitation, and falls. Use of a locally administered liposomal bupivacaine could decrease the need for additional medications for pain control in addition to decreased mental stress for patients in this unfamiliar situation, thus resulting in decreased episodes of delirium. The investigators will assess delirium utilizing Confusion Assessment Method (CAM) scores in the post-operative period at regularly scheduled intervals and compare average scores between the treatment / standard of care group. Hypothesis: The investigators hypothesize that total episodes of delirium will be decreased in the liposomal bupivacaine group.
3. Determine if Exparel is cost-effective in hip fracture patients. The costs associated with increased narcotic usage, prolonged stay, resources, and complications can be significant. The use of liposomal bupivacaine may lead to decreased resource utilization to care for hip fractures. The investigators will conduct an economic analysis evaluating total inpatient hospitalization costs including costs associated with length of stay, medication requirements, and resources associated with consultations and diagnostic evaluations. These costs will be compared against the cost of Exparel administration to evaluate the net cost effect of the intervention. Hypothesis: The investigators hypothesize that the net cost of inpatient care will be decreased when compared to standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 or older
* Sustaining either an OTA/AO type 31A or 31B fracture undergoing ORIF or hemiarthroplasty
* Able to consent
* Isolated injury

Exclusion Criteria:

* OTA/AO 31B1 (Impacted/slightly displaced)
* Baseline dementia or cognitive deficit
* Inability to consent
* Chronic Opioid use
* End stage liver disease with Model for End-Stage Liver Disease (MELD) greater than 20.
* End stage renal disease as defined by patients requiring hemodialysis at least twice weekly
* Polytrauma, defined as: concurrent upper or lower extremity fracture, pelvis fracture, spine fracture, rib fractures, or facial fractures, Blunt chest or abdominal trauma resulting in diagnosed organ injury, Head trauma resulting in intracranial bleed or diagnosed concussion
* Allergy to amide-type local anesthetics
* Prisoners (unlikely to be accessible for follow-up)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Swart, MD, Principal Investigator — UMass Memorial Health; Paul Matuszewski, MD, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - University of Kentucky, Lexington, Kentucky
  - UMass Memorial Medical Center, Worcester, Massachusetts

REFERENCES:
- [Background] Brauer CA, Coca-Perraillon M, Cutler DM, Rosen AB. Incidence and mortality of hip fractures in the United States. JAMA. 2009 Oct 14;302(14):1573-9. doi: 10.1001/jama.2009.1462. PMID 19826027
- [Background] Burge R, Dawson-Hughes B, Solomon DH, Wong JB, King A, Tosteson A. Incidence and economic burden of osteoporosis-related fractures in the United States, 2005-2025. J Bone Miner Res. 2007 Mar;22(3):465-75. doi: 10.1359/jbmr.061113. PMID 17144789
- [Background] Sanzone AG. Current Challenges in Pain Management in Hip Fracture Patients. J Orthop Trauma. 2016 May;30 Suppl 1:S1-5. doi: 10.1097/BOT.0000000000000562. PMID 27101319
- [Background] Koval KJ, Zuckerman JD. Hip Fractures: I. Overview and Evaluation and Treatment of Femoral-Neck Fractures. J Am Acad Orthop Surg. 1994 May;2(3):141-149. doi: 10.5435/00124635-199405000-00002. PMID 10709002
- [Background] Koval KJ, Zuckerman JD. Hip Fractures: II. Evaluation and Treatment of Intertrochanteric Fractures. J Am Acad Orthop Surg. 1994 May;2(3):150-156. doi: 10.5435/00124635-199405000-00003. PMID 10709003
- [Background] Chau DL, Walker V, Pai L, Cho LM. Opiates and elderly: use and side effects. Clin Interv Aging. 2008;3(2):273-8. doi: 10.2147/cia.s1847. PMID 18686750
- [Background] Lonner JH, Scuderi GR, Lieberman JR. Potential utility of liposome bupivacaine in orthopedic surgery. Am J Orthop (Belle Mead NJ). 2015 Mar;44(3):111-7. PMID 25750943
- [Background] Berend ME, Berend KR, Lombardi AV Jr. Advances in pain management: game changers in knee arthroplasty. Bone Joint J. 2014 Nov;96-B(11 Supple A):7-9. doi: 10.1302/0301-620X.96B11.34514. PMID 25381400
- [Background] Ma J, Zhang W, Yao S. Liposomal bupivacaine infiltration versus femoral nerve block for pain control in total knee arthroplasty: A systematic review and meta-analysis. Int J Surg. 2016 Dec;36(Pt A):44-55. doi: 10.1016/j.ijsu.2016.10.007. Epub 2016 Oct 11. PMID 27742564
- [Background] Cherian JJ, Muzaffar A, Barrington JW, Elmallah RD, Chughtai M, Mistry JB, Mont MA. Liposomal Bupivacaine in Total Knee Arthroplasty for Better Postoperative Analgesic Outcome and Economic Benefits. J Knee Surg. 2016 Jul;29(5):e2. doi: 10.1055/s-0036-1584270. Epub 2016 Jun 10. No abstract available. PMID 27285179
- [Background] Chughtai M, Cherian JJ, Mistry JB, Elmallah RD, Bennett A, Mont MA. Liposomal Bupivacaine Suspension Can Reduce Lengths of Stay and Improve Discharge Status of Patients Undergoing Total Knee Arthroplasty. J Knee Surg. 2016 Apr;29(3):224-7. doi: 10.1055/s-0036-1571431. Epub 2016 Feb 2. PMID 26838971
- [Background] Surdam JW, Licini DJ, Baynes NT, Arce BR. The use of exparel (liposomal bupivacaine) to manage postoperative pain in unilateral total knee arthroplasty patients. J Arthroplasty. 2015 Feb;30(2):325-9. doi: 10.1016/j.arth.2014.09.004. Epub 2014 Sep 16. PMID 25282071
- [Background] Zuckerman JD. Hip fracture. N Engl J Med. 1996 Jun 6;334(23):1519-25. doi: 10.1056/NEJM199606063342307. No abstract available. PMID 8618608
- [Background] Menzies IB, Mendelson DA, Kates SL, Friedman SM. The impact of comorbidity on perioperative outcomes of hip fractures in a geriatric fracture model. Geriatr Orthop Surg Rehabil. 2012 Sep;3(3):129-34. doi: 10.1177/2151458512463392. PMID 23569706
- [Background] Zywiel MG, Hurley RT, Perruccio AV, Hancock-Howard RL, Coyte PC, Rampersaud YR. Health economic implications of perioperative delirium in older patients after surgery for a fragility hip fracture. J Bone Joint Surg Am. 2015 May 20;97(10):829-36. doi: 10.2106/JBJS.N.00724. PMID 25995494
- [Background] Marcantonio ER, Flacker JM, Wright RJ, Resnick NM. Reducing delirium after hip fracture: a randomized trial. J Am Geriatr Soc. 2001 May;49(5):516-22. doi: 10.1046/j.1532-5415.2001.49108.x. PMID 11380742
- [Background] Ma TT, Wang YH, Jiang YF, Peng CB, Yan C, Liu ZG, Xu WX. Liposomal bupivacaine versus traditional bupivacaine for pain control after total hip arthroplasty: A meta-analysis. Medicine (Baltimore). 2017 Jun;96(25):e7190. doi: 10.1097/MD.0000000000007190. PMID 28640101
- [Background] Asche CV, Ren J, Kim M, Gordon K, McWhirter M, Kirkness CS, Maurer BT. Local infiltration for postsurgical analgesia following total hip arthroplasty: a comparison of liposomal bupivacaine to traditional bupivacaine. Curr Med Res Opin. 2017 Jul;33(7):1283-1290. doi: 10.1080/03007995.2017.1314262. Epub 2017 Apr 28. PMID 28375752
- [Background] McGraw-Tatum MA, Groover MT, George NE, Urse JS, Heh V. A Prospective, Randomized Trial Comparing Liposomal Bupivacaine vs Fascia Iliaca Compartment Block for Postoperative Pain Control in Total Hip Arthroplasty. J Arthroplasty. 2017 Jul;32(7):2181-2185. doi: 10.1016/j.arth.2017.02.019. Epub 2017 Feb 16. PMID 28318860
- [Background] Yu SW, Szulc AL, Walton SL, Davidovitch RI, Bosco JA, Iorio R. Liposomal Bupivacaine as an Adjunct to Postoperative Pain Control in Total Hip Arthroplasty. J Arthroplasty. 2016 Jul;31(7):1510-5. doi: 10.1016/j.arth.2016.01.004. Epub 2016 Jan 21. PMID 26872584
- [Background] Domb BG, Gupta A, Hammarstedt JE, Stake CE, Sharp K, Redmond JM. The effect of liposomal bupivacaine injection during total hip arthroplasty: a controlled cohort study. BMC Musculoskelet Disord. 2014 Sep 24;15:310. doi: 10.1186/1471-2474-15-310. PMID 25248686
- [Background] Barrington JW, Olugbode O, Lovald S, Ong K, Watson H, Emerson RH Jr. Liposomal Bupivacaine: A Comparative Study of More Than 1000 Total Joint Arthroplasty Cases. Orthop Clin North Am. 2015 Oct;46(4):469-77. doi: 10.1016/j.ocl.2015.06.003. Epub 2015 Aug 6. PMID 26410636
- [Background] Cherian JJ, Barrington J, Elmallah RK, Chughtai M, Mistry JB, Mont MA. Liposomal Bupivacaine Suspension, Can Reduce Length of Stay and Improve Discharge Status of Patients Undergoing Total Hip Arthroplasty. Surg Technol Int. 2015 Nov;27:235-9. PMID 26680403
- [Background] Hutchinson HL. Local infiltration of liposome bupivacaine in orthopedic trauma patients: case-based reviews. Am J Orthop (Belle Mead NJ). 2014 Oct;43(10 Suppl):S13-6. PMID 25303455
- [Background] Herbst SA. Local infiltration of liposome bupivacaine in foot and ankle surgery: case-based reviews. Am J Orthop (Belle Mead NJ). 2014 Oct;43(10 Suppl):S10-2. PMID 25303454
- [Background] Morrison RS, Dickman E, Hwang U, Akhtar S, Ferguson T, Huang J, Jeng CL, Nelson BP, Rosenblatt MA, Silverstein JH, Strayer RJ, Torrillo TM, Todd KH. Regional Nerve Blocks Improve Pain and Functional Outcomes in Hip Fracture: A Randomized Controlled Trial. J Am Geriatr Soc. 2016 Dec;64(12):2433-2439. doi: 10.1111/jgs.14386. Epub 2016 Oct 27. PMID 27787895
- [Background] Yokomizo JE, Simon SS, Bottino CM. Cognitive screening for dementia in primary care: a systematic review. Int Psychogeriatr. 2014 Nov;26(11):1783-804. doi: 10.1017/S1041610214001082. Epub 2014 Jul 15. PMID 25023857
- [Background] Wei LA, Fearing MA, Sternberg EJ, Inouye SK. The Confusion Assessment Method: a systematic review of current usage. J Am Geriatr Soc. 2008 May;56(5):823-30. doi: 10.1111/j.1532-5415.2008.01674.x. Epub 2008 Apr 1. PMID 18384586
- [Background] White PF, Issioui T, Skrivanek GD, Early JS, Wakefield C. The use of a continuous popliteal sciatic nerve block after surgery involving the foot and ankle: does it improve the quality of recovery? Anesth Analg. 2003 Nov;97(5):1303-1309. doi: 10.1213/01.ANE.0000082242.84015.D4. PMID 14570643
- [Background] Busch CA, Shore BJ, Bhandari R, Ganapathy S, MacDonald SJ, Bourne RB, Rorabeck CH, McCalden RW. Efficacy of periarticular multimodal drug injection in total knee arthroplasty. A randomized trial. J Bone Joint Surg Am. 2006 May;88(5):959-63. doi: 10.2106/JBJS.E.00344. PMID 16651569
- [Background] Ng FY, Ng JK, Chiu KY, Yan CH, Chan CW. Multimodal periarticular injection vs continuous femoral nerve block after total knee arthroplasty: a prospective, crossover, randomized clinical trial. J Arthroplasty. 2012 Jun;27(6):1234-8. doi: 10.1016/j.arth.2011.12.021. Epub 2012 Feb 8. PMID 22325963
- [Derived] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exparel (Liposomal Bupivacaine) | Saline Control
Started | 27 | 28
Completed | 25 | 28
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exparel (Liposomal Bupivacaine) | Saline Control | Total
Number analyzed (Participants) | 27 | 28 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 76 (8.6) | 77 (9.2) | 76 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 7 | 8 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 27 | 28 | 55

OUTCOME MEASURES:

1. Primary Outcome: Opiate Requirements
Description: Morphine meq given
Time Frame: 72 hours
Measure: Mean (95% Confidence Interval); unit: Morphine mEq
Arm/Group | Exparel (Liposomal Bupivacaine) | Saline Control
Number analyzed (Participants) | 25 | 28
Morphine mEq | 52.5 [30.21 to 74.75] | 65.39 [45.68 to 85.10]

ADVERSE EVENTS:
Time Frame: 3 months
Description: Patients were actively screened for a list of complications daily during their admission and at their 2 and 6 week follow up appointments.
Arm/Group | Exparel (Liposomal Bupivacaine) | Saline Control
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/27 | 1/28
Other Adverse Events (participants affected / at risk) | 0/27 | 0/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exparel (Liposomal Bupivacaine) (N=27) | Saline Control (N=28)
Infection (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/58/NCT03289858/Prot_003.pdf
  • Statistical Analysis Plan (2017-08-27): https://cdn.clinicaltrials.gov/large-docs/58/NCT03289858/SAP_004.pdf